CLINICAL TRIAL: NCT03818503
Title: E²-RADIatE: EORTC-ESTRO RADiotherapy InfrAstrucTure for Europe
Acronym: E²-RADIatE
Status: Recruiting | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1811
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OligoCare: Patients with oligometastatic disease treated with radical radiotherapy
- ReCare: Patients treated with high-dose Re-irradiation

SUMMARY:
The primary objective is the collection of real-world data of cancer patients treated with radiotherapy, to support radiotherapy research and to provide evidence of the role of radiation oncology in a multidisciplinary approach. This is an open ended prospective non-interventional non-therapeutic multi-cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cancer.
* Written informed consent for E²-RADIatE according to applicable legal and ethical requirements
* Planned use of radiotherapy
* Eligibility of the patient confirmed for at least one cohort confirmed
* Patients of 12 years and older

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with various tumor types planned to be treated with radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with radiotherapy enrolled in the program | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years
Loco-regional control | 5 years
Distant metastasis free survival | 5 years
Overall survival | 5 years
Incidence of adverse events related to radiotherapy | 5 years

CONTACTS AND LOCATIONS:
Locations (77):
- Austria (3):
  - Medical University of Graz - Radio-oncology, Graz
  - Ordensklinikum Linz-Barmherzige Schwestern, Linz
  - Universitaetskliniken der Uni Wien - Universitaetsklinikum Wien - AKH unikliniken, Vienna
- Belgium (11):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Sint-Lucas & Volkskliniek, Ghent
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - C.H.U. Sart-Tilman, Liège
  - CHU Site Sainte-Elisabeth-UCL Namur, Namur
  - AZ Turnhout - Campus Sint Elisabeth, Turnhout
  - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
- University Hospital Hradec Kralove, Hradec Králové, Czechia
- Clinique Pasteur-Lanroze (1174), Brest, France
- Germany (5):
  - Universitaetsklinikum Aachen AOR - Medizinische Fakultaet der RWTH, Aachen
  - Klinikum Bayreuth Gmbh, Bayreuth
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Ludwig-Maximilians-Universitaet Muenchen - Campus Grosshadern, München
- Ireland (3):
  - St Luke Hospital & SLRON - SLRON - St. Luke'S Hospital Rathgar, Dublin
  - Beacon Hospital, Dublin
  - University Hospital Galway, Galway
- Sheba Medical Center Tel Hashomer, Ramat Gan, Israel
- Italy (16):
  - Ente Ecclesiastico Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - USL Toscana South East, Ospedale S. Donato, Arezzo
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Univ. of Florence -Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Sacro Cuore Hospital, Negrar
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Centro Nazionale di Adroterapia Oncoloica par il trattamento dei tumori, Pavia
  - San Maria della Misericordia Hospital, Perugia
  - Policlinico Universitario Campus Bio-Medico- Oncology Center, Roma
  - Fondazione Policlinico Universitario A. Gemelli - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino - Universita Di Torino - San Giovanni Battista, Torino
- Netherlands (4):
  - Stichting Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Groningen
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
  - Radiotherapiegroep Arnhem, Nijmegen
- Poland (3):
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Kliniki Neuroradiochirurgii Sp. z o.o.-Radomskie Centrum Onkologii, Radom
  - Maria Sklodowska-Curie Memorial Cancer Centre - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- The Institute Of Oncology, Ljubljana, Slovenia
- Spain (15):
  - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona
  - Hospital Universitari Vall d'Hebron -Vall d'Hebron Institut Oncologia, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Santa Lucia, Cartagena
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospitales HM Sanchinarro-CIOCC, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario de Salamanca (430), Salamanca
  - Hospital Consorci Sanitari De Terrassa, Terrassa
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
- Switzerland (6):
  - Inselspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
  - Reseau Hospitalier Neuchatelois - RHNe - La Chaux de Fonds, La Chaux-de-Fonds
  - Hopital du Valais - Hopital de Sion, Sion
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (7):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - Velindre NHS Trust - Velindre Cancer Centre, Cardiff
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - The Christie NHS Foundation trust - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge cancer Center NHS foundation Trust - Clatterbridge Cancer Center - Wirral, Metropolitan Borough of Wirral
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield
  - Somerset NHS Foundation Trust-Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christ SM, Alongi F, Ricardi U, Scorsetti M, Livi L, Balermpas P, Lievens Y, Braam P, Jereczek-Fossa BA, Stellamans K, Ratosa I, Widder J, Peulen H, Dirix P, Bral S, Ramella S, Hemmatazad H, Khanfir K, Geets X, Jeene P, Zilli T, Fournier B, Ivaldi GB, Clementel E, Fortpied C, Oppong FB, Ost P, Guckenberger M. Cancer-specific dose and fractionation schedules in stereotactic body radiotherapy for oligometastatic disease: An interim analysis of the EORTC-ESTRO E2-RADIatE OligoCare study. Radiother Oncol. 2024 Jun;195:110235. doi: 10.1016/j.radonc.2024.110235. Epub 2024 Mar 19. PMID 38508239
- [Derived] Nieder C, Willmann J, Andratschke NH. Prospective randomized clinical studies involving reirradiation: update of a systematic review. Strahlenther Onkol. 2023 Sep;199(9):787-797. doi: 10.1007/s00066-023-02118-1. Epub 2023 Jul 27. PMID 37500926